CLINICAL TRIAL: NCT05217498
Title: A Selective Adenosine 2a Antagonist to Enhance Training-related Gains in Walking Function for Persons With Chronic, Incomplete Spinal Cord Injury
Brief Title: Combining Low Oxygen Therapy and an Adenosine A2a Receptor Antagonist to Improve Functional Mobility After Spinal Cord Injury
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Randy Trumbower, PT, PhD (Other)
Responsible Party: Sponsor-Investigator, Randy Trumbower, PT, PhD, Assistant Professor, Spaulding Rehabilitation Hospital
Organization: Spaulding Rehabilitation Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018A004512
Record Dates: First submitted 2022-01-11; First posted 2022-02-01 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Myelopathy
Keywords: spinal cord injury; walking; motor control; istradefylline; adenosine; strength
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases | interventions — istradefylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Istradefylline+low oxygen training (Experimental): Drug: Nourianz Other Names: KW6002, Istradefylline
  Participants enrolled in this study arm will ingest a 20mg tablet/day containing istradefylline starting 14 days prior to the first low oxygen therapy and continuing for 14 additional days. Participants will consume a total of 28 istradefylline tablets.
  Other: low oxygen training Other Names: therapeutic intermittent hypoxia, acute intermittent hypoxia
  Participants will breathe 15 episodes/session of acute low oxygen via an automated air generator system (4 sessions/week x 2 weeks). During the 90-second episodes of low oxygen, air concentrations will be continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.10±0.02 (hypoxia) with 60-second room-air intervals (FIO2 0.21±0.02).
  Throughout experimentation, blood pressure, respiratory rate, and heart rate will be monitored. We also will assess for changes in sleep quality and pain level.
  Interventions: Drug: Istradefylline; Device: low oxygen therapy
- Placebo+low oxygen training (Active Comparator): This is a placebo counterpart to the istradefylline drug.
  Participants enrolled in this study arm will ingest a 20mg placebo tablet/day containing dextrose starting 14 days prior to the first low oxygen therapy (LOT) and continuing for 14 additional days. Participants will consume a total of 28 placebo tablets.
  Other: low oxygen training Other Names: therapeutic intermittent hypoxia, acute intermittent hypoxia
  Participants will breathe 15 episodes/session of acute low oxygen via an automated air generator system (4 sessions/week x 2 weeks). During the 90-second episodes of low oxygen, air concentrations will be continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.10±0.02 (hypoxia) with 60-second room-air intervals (FIO2 0.21±0.02).
  Throughout experimentation, blood pressure, respiratory rate, and heart rate will be monitored. We also will assess for changes in sleep quality and pain level.
  Interventions: Device: low oxygen therapy
- Istradefylline+SHAM (Active Comparator): Drug: Nourianz Other Names: KW6002, Istradefylline
  This is a SHAM counterpart to low oxygen therapy.
  Participants enrolled in this study arm will ingest a 20mg tablet/day containing istradefylline starting 14 days prior to the first SHAM therapy and continuing for 14 additional days. Participants will consume a total of 28 istradefylline tablets.
  Participants will breathe 15 episodes/session of SHAM via an automated air generator system (4 sessions/week x 2 weeks). The system will fill reservoir bags attached to a non-rebreathing face mask. During the 90-second episodes of SHAM, air concentrations will be continuously monitored to ensure delivery of FIO2 (fraction of inspired oxygen) = 0.21±0.02 (normoxia) with 60-second room-air intervals (FIO2 0.21±0.02).
  Throughout experimentation, blood pressure, respiratory rate, and heart rate will be monitored. We also will assess for changes in sleep quality and pain level.
  Interventions: Drug: Istradefylline

INTERVENTIONS:
Drug: Istradefylline — Consume 20mg tablet of istradefylline for 28 consecutive days.
  Other Names: KW6002; Nourianz
  Arms: Istradefylline+SHAM; Istradefylline+low oxygen training
Device: low oxygen therapy — Breath intermittent low oxygen 4 days/week over 2 consecutive weeks. Intermittent low oxygen consists of 15, 90-second episodes of breathing low oxygen at 10% oxygen with 60-second intervals at 21% oxygen.
  Other Names: acute intermittent hypoxia
  Arms: Istradefylline+low oxygen training; Placebo+low oxygen training

SUMMARY:
Breathing brief, moderate bouts of low oxygen trigger (low oxygen therapy, LOT) spinal plasticity (the ability of the nervous system to strengthen neural pathways based on new experiences), and improve walking after spinal cord injury (SCI). The greatest improvements in walking ability occur when LOT is administered prior to skill-based walking practice (WALK). However, the enduring benefits of LOT on walking recovery may be undermined by the accumulation of LOT-induced increase in extracellular adenosine. The goal of the study is to understand the extent to which istradefylline (adenosine 2a receptor antagonist) may limit the competing mechanisms of adenosine on LOT-induced walking recovery following SCI.

DETAILED DESCRIPTION:
This randomized, placebo-controlled clinical trial will examine the efficacy of a selective adenosine 2a antagonist (istradefylline) to enhance the beneficial effects of LOT-related gains on overground walking performance after spinal cord injury (SCI).

Participants will be randomly assigned to a combinatorial intervention: istradefylline+LOT, placebo+LOT, istradefylline+SHAM. Participants will be asked to avoid caffeine-containing substances for 48 hrs (> 5* half-life of ~7 hrs) before the start of the study. They also will refrain from consuming caffeine during the 4-week combinatorial intervention.

Participants enrolled in istradefylline+AIH will receive 20mg of istradefylline orally for 28 consecutive days. After 14 days of istradefylline treatment, the participants will receive 2 weeks (4 sessions/week) of LOT prior to 45min of skill-based walking practice (WALK) within the INSPIRE Lab. A single session of LOT will consist of 15 episodes of breathing 90s low levels of oxygen (10% O2) with 60s intervals at room air (21% O2).

Participants enrolled in istradefylline+SHAM will receive 20mg of istradefylline orally for 28 consecutive days. After 14 days of istradefylline treatment, the participants will receive 2 weeks (4 sessions/week) of SHAM therapy prior to 45min of skill-based walking practice (WALK) within the INSPIRE Lab. A single session of SHAM therapy will consist of 15 episodes of breathing 90s of normal levels of oxygen (21% O2) with 60s intervals at room air (21% O2).

Participants enrolled in placebo+AIH will receive 20mg of placebo (dextrose) treatment orally for 28 consecutive days. After 14 days of placebo treatment, the participants will receive 2 weeks (4 sessions/week) of LOT prior to 45min of skill-based walking practice (WALK) within the INSPIRE Lab. A single session of LOT will consist of 15 episodes of breathing 90s low levels of oxygen (10% O2) with 60s intervals at room air (21% O2).

Blood samples will be collected at baseline, and at the end of week 2, week 4 to assess for potential confounding effects of systemic inflammation and caffeine on responsiveness to the combinatorial interventions.

The study will assess functional outcomes, vital signs, and symptoms before and after each intervention. For our primary outcome measure, the study will assess walking speed (10-meter walk test, 10MWT) relative to baseline at the end of day 5 (D5), and 8 (F1) and 14 days (F2) post-treatment. This study also will assess leg strength, walking distance, and coordination on D5, F1, and F2 as secondary outcome measures. A linear mixed model will be used to compare differences in 10MWT with treatment and time as main effects and participants as random effects. This study will follow the Consolidated Standards of Reporting Trials.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 and 75 years (the latter to reduce the likelihood of heart disease) medical clearance to participate
2. lesion at or below C2 and above T12 with non-progressive etiology
3. classified as motor-incomplete with visible volitional leg movement
4. injury greater than 12 months
5. ability to advance one step overground without human assistance

Exclusion Criteria:

1. Concurrent severe medical illness (i.e., infection, cardiovascular disease, ossification, recurrent autonomic dysreflexia, unhealed decubiti, and history of pulmonary complications)
2. Pregnant women because of the unknown effects of AIH on pregnant women and fetus
3. History of seizures, brain injury, and/or epilepsy
4. Undergoing concurrent physical therapy
5. Diabetes
6. Cirrhosis Caffeine and/or NSAID allergies or intolerances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-09-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-Treatment Walking Speed | within 5 days of first treatment
  Pre-Treatment Walking Speed; 10MWT (time, seconds)
Walking Speed Post-Treatment 1 | within 1 day after last treatment
  Post-Treatment Walking Speed; 10MWT (time, seconds)
Walking Speed Post-Treatment 2 | between 7-10 days after Post-Treatment 1
  Post-Treatment Walking Speed; 10MWT (time, seconds)
Walking Speed Post-Treatment 3 | between 17-20 days after Post-Treatment 1
  Post-Treatment 10MWT (time, seconds)

SECONDARY OUTCOMES:
Pre-Treatment Walking Distance | within 5 days of first treatment
  Pre-Treatment 6MWT (distance, meters)
Walking Distance Post-Treatment 1 | within 1 day after last treatment
  Post-Treatment 6MWT (distance, meters)
Walking Distance Post-Treatment 2 | between 7-10 days after Post-Treatment 1
  Post-Treatment 6MWT (distance, meters)
Walking Distance Post-Treatment 3 | between 17-20 days after Post-Treatment 1
  Post-Treatment 6MWT (distance, meters)
Pre-Treatment Timed Up-and-Go Test | within 5 days of first treatment
  Pre-Treatment TUG (walking balance)
Timed Up-and-Go Test Post-Treatment 1 | within 1 day after last treatment
  Post-Treatment TUG (walking balance)
Timed Up-and-Go Test Post-Treatment 2 | between 7-10 days after Post-Treatment 1
  Post-Treatment TUG (walking balance)
Timed Up-and-Go Test Post-Treatment 3 | between 17-20 days after Post-Treatment 1
  Post-Treatment TUG (walking balance)
Pre-treatment Ankle Strength | within 5 days of first treatment
  Pre-Treatment Plantarflexion Torque (strength, torque)
Ankle Strength Post-Treatment 1 | within 1 day after last treatment
  Post-Treatment Plantarflexion Torque (strength, torque)
Ankle Strength Post-Treatment 2 | between 7-10 days after Post-Treatment 1
  Post-Treatment Plantarflexion Torque (strength, torque)
Ankle Strength Post-Treatment 3 | between 17-20 days after Post-Treatment 1
  Post-Treatment Plantarflexion Torque (strength, torque)

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Trumbower, PT, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Tan AQ, Papadopoulos JM, Corsten AN, Trumbower RD. An automated pressure-swing absorption system to administer low oxygen therapy for persons with spinal cord injury. Exp Neurol. 2020 Nov;333:113408. doi: 10.1016/j.expneurol.2020.113408. Epub 2020 Jul 17. PMID 32682613
- [Background] Tan AQ, Barth S, Trumbower RD. Acute intermittent hypoxia as a potential adjuvant to improve walking following spinal cord injury: evidence, challenges, and future directions. Curr Phys Med Rehabil Rep. 2020 Sep;8(3):188-198. doi: 10.1007/s40141-020-00270-8. Epub 2020 Jun 24. PMID 33738145
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Trumbower RD, Hayes HB, Mitchell GS, Wolf SL, Stahl VA. Effects of acute intermittent hypoxia on hand use after spinal cord trauma: A preliminary study. Neurology. 2017 Oct 31;89(18):1904-1907. doi: 10.1212/WNL.0000000000004596. Epub 2017 Sep 29. PMID 28972191
- [Background] Vivodtzev I, Tan AQ, Hermann M, Jayaraman A, Stahl V, Rymer WZ, Mitchell GS, Hayes HB, Trumbower RD. Mild to Moderate Sleep Apnea Is Linked to Hypoxia-induced Motor Recovery after Spinal Cord Injury. Am J Respir Crit Care Med. 2020 Sep 15;202(6):887-890. doi: 10.1164/rccm.202002-0245LE. No abstract available. PMID 32369393
- [Background] Tan AQ, Sohn WJ, Naidu A, Trumbower RD. Daily acute intermittent hypoxia combined with walking practice enhances walking performance but not intralimb motor coordination in persons with chronic incomplete spinal cord injury. Exp Neurol. 2021 Jun;340:113669. doi: 10.1016/j.expneurol.2021.113669. Epub 2021 Feb 27. PMID 33647273
- See also: Research Lab Website — https://www.inspire-lab.org